CLINICAL TRIAL: NCT03583177
Title: Study of Muscle Wasting Mechanisms and Biomarkers in Hemodialysis Patient
Brief Title: Muscle Wasting in Hemodialysis Patient
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-397; 2008-A00479-46 (Other: 2008-A00479-46)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Muscle Atrophy in Lung Cancer and Hemodialysed Patients
Keywords: Proteolysis; Muscle; Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers
  Interventions: Diagnostic Test: No intervention
- cancer patients
  Interventions: Diagnostic Test: No intervention
- undergoing chronic hemodialysis patients
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Muscle wasting is present in almost 50% of patients treated with chronic hemodialysis. It is associated with an increased risk of death (particularly from cardiovascular causes) and compromises quality of life (loss of autonomy and fatigue). The mechanisms leading to muscle wasting in chronic kidney disease have been the subject of several studies in animals. These have highlighted the role of the ubiquitin-proteasome system (UPS). Activation of UPS during chronic kidney disease is multifactorial. It is the result of resistance to the action of insulin/IGF1, metabolic acidosis, low grade prolonged inflammation and increased production of myostatin. To date few studies have been conducted in humans.

The investigators want to identify blood markers related to muscle protein breakdown in patients undergoing hemodialysis. In parallel, the investigators want to adress the mechanisms involved in muscle proteolysis. In addition, the investigators want to identify the proteins degraded and the ubiquitination enzymes (E2/E3 couples) specifically involved in muscle loss during hemodialysis.

Muscle biopsies and blood sample will beperformed during scheduled surgeries in healthy volunteers (negative control), cancer patients (positive control) or undergoing chronic hemodialysis. RNA seq analysis will be performed in blood samples and proteomic mass spectrometry analysis for establishing a specific profile between muscle and blood markers. A limited subset of blood markers common to cancer and hemodialysis atrophying muscles will be used for elaborating a chip dedicated to early detect an atrophying process.

Thus, the investigators will first design a diagnostic tool for detecting non-invasively muscle protein breakdown before the onset of muscle atrophy. This will enable early and efficient nutritional counter-measures.

DETAILED DESCRIPTION:
Hypothesis Measuring urinary 3-methylhistidine is a simple tool to assess proteolysis in clinical practice. However it is not totally specific of muscle proteolysis because it may reflect an intestinal catabolism. Moreover, its dosage cannot be used in patients with renal impairment especially in case of anuria. Apart from achieving muscle biopsy or measuring the overall kinetics of proteins it does not yet exist simple and reproducible diagnostic tool for measuring muscle proteolysis. With the present study, the investigators expect to identify in the blood of patients a particular transcriptomic profile related to the activation of muscle proteolysis, including increased proinflammatory cytokine transcripts.

Rodent models of CKD were used to identify major proteolytic system and signal pathway implicated in muscle wasting caused by uremia. These finding needs to be confirmed in humans studies. Also, other actors of muscle atrophy could be identified in humans. Notably, so far, few studies have been performed in order to determine which E2 are involved in muscle atrophy, and to knowledge of the investigators no one in CKD. Finally, data on muscle proteasome substrates are limited since only actin was clearly identified in humans by the team. The investigators expect an activation of the proteasome system with an increase in the expression of enzymes E2s, E3s including MURF1 and MAFbx and proteasome subunit in patients treated with hemodialysis. The investigators could also observe an activation of caspase system which is thought to work in concert with the UPS.

Materials and methods 2.1. Population The experiments will be performed using blood sample and human muscle biopsies obtained during programmed orthopedic surgery (negative control), cancer (positive control) and hemodialysis patients. This translational research program has already been accepted (DGS 2008-A00479-46) and inclusion of patients already started. A maximum of 15 patients per group will be included. Inclusion and exclusion criteria were set-up according to the objectives (absence of any pathology for controls, etc.) and the legislation (written consent, etc.). Thirty-two patients have already been included so far, and biopsies are stored in liquid nitrogen. Blood samples are collected just before surgery using Paxgene RNA tubes and stored following the manufacturer's instructions until analysis.

2.2. Blood sample Total RNA will be extracted from blood using Paxgene RNA Extraction kit and analysed by RNAseq 2.3. Muscle biopsies 2.3.1. Transcriptomic analysis Total RNA will be extracted from human muscle biopsies using commercial kits. The investigators will first verify that known muscles markers are up-regulated in cancer patient biopsies (positive controls) and address their levels in muscle biopsies from hemodialysis patients. We will thus perform qRT-PCR UBE2B, UBE2D2, MaFbx, MuRF1, Ozz, ASB2, E4B, Nedd4, Mdm2 and 26S proteasome subunits.

2.3.2. Proteomic analysis Proteomic analysis will be performed usin shot gun spectrometry analysis

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* with either newly diagnosed lung cancer (for whom surgical resection was programmed by thoracotomy) or patients with end-stage renal failure treated for at least 6 months by hemodialysis and necessitating femoral bypass revascularization.
* The control group patients required hip replacement for osteoarthritis.

Exclusion Criteria:

* acute or chronic infections,
* diabetes mellitus,
* corticosteroid or hormone therapy or
* pregnancy.
* Glomerular filtration rate < 90 mL/min for LC and CT patients
* active neoplasia in patients of the HD and CT groups
* CRP > 3 mg/L in for CT patients

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Both female and male participants from18 years old to 75 years old are being studied. Those 40 patients are either affected by cancer or hemodialysis volunteer, or constitute group control.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Transcriptomic analysis of total blood sample | From July 2009 to July 2011
  Total RNA will be extracted from blood using Paxgene RNA Extraction kit and analysed by RNAseq and a comparison made between patients and control.
To find biomarkers of muscle atrophy | From July 2009 to July 2011
  1. To confirm the implication of UPS in muscular proteolysis of IRCH patients by the detection of an increasing of ARNm, except ubiquitin, implicated in the quantitative RT-PCR system and by the identification of substrates.
  2. To locate on the proteins that have to be deteriorated, the sites used by the UPS to fix polyubiquitin chains.

SECONDARY OUTCOMES:
Transcriptomic analysis | From July 2009 to July 2011
  Total RNA will be extracted from human muscle biopsies using commercial kits. We will first verify that known muscles markers are up-regulated in cancer patient biopsies (positive controls) and address their levels in muscle biopsies from hemodialysis patients. We will thus perform qRT-PCR UBE2B, UBE2D2, MaFbx, MuRF1, Ozz, ASB2, E4B, Nedd4, Mdm2 and 26S proteasome subunits.
Proteomic analysis in muscle biopsies for identification of cachexia mechanism | From July 2009 to July 2011
  Proteomic analysis will be performed usin shot gun spectrometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Julien ANIORT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France